CLINICAL TRIAL: NCT02829723
Title: A Phase I/II, Open-label, Multi-center Study of the Safety and Efficacy of BLZ945 as Single Agent and in Combination With PDR001 in Adults Patients With Advanced Solid Tumors
Brief Title: A Study of BLZ945 Single Agent or BLZ945 in Combination With PDR001 in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBLZ945X2101; 2015-005806-12 (EudraCT Number)
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Results first posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-12

CONDITIONS: Advanced Solid Tumors
Keywords: Phase I/II; BLZ945; PDR001; CSF-1R; PD-1; advanced solid tumors; glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — 4-(2-(2-hydroxycyclohexylamino)benzothiazol-6-yloxy)pyridine-2-carboxylic acid methylamide; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BLZ945 single agent (Experimental): BLZ945 administered as single agent
  Interventions: Drug: BLZ945
- BLZ945 + PDR001 (Experimental): BLZ945 administered in combination with PDR001
  Interventions: Drug: BLZ945; Drug: PDR001

INTERVENTIONS:
Drug: BLZ945 — BLZ945 administered orally as a capsule. Up to five alternative dosing schedules were evaluated: once per day (QD) 7 days on/7 days off (i.e., administer BLZ945 for 7 days and suspend for 7 days), QD 4 days on/10 days off, twice per day (BID) 4 days on/10 days off, once weekly (Q1W) QD and Q1W BID.
  Each cycle consisted of 28 days.
Drug: PDR001 — PDR001 400 mg administered via intravenous (i.v.) infusion every 4 weeks (Q4W)
  Other Names: spartalizumab
  Arms: BLZ945 + PDR001

SUMMARY:
The purpose of this first-in-human (FIH) study of BLZ945 given as a single agent or in combination with PDR001 was to characterize the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and anti-tumor activity of BLZ945, administered orally, as a single agent or in combination with PDR001, administered intravenously (i.v.) in adult patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study was a first in human, open-label, multi-center phase I/II study which consisted of a phase I dose escalation part of BLZ945 as single agent, and of BLZ945 in combination with PDR001, where alternative dosing regimens of BLZ945 were evaluated. The escalation was guided by a Bayesian logistic regression model with overdose control. Once the maximum tolerated dose (MTD) / recommended phase 2 dose (RP2D) for BLZ945 as single agent was established, a phase II part could commence, should signs of antitumor activity had been seen during the phase I. Once the MTD/RP2D for BLZ945 in combination with PDR001 was established, a phase II part could commence.

Phase I part of the study involved patients with advanced solid tumors, including patients with recurrent glioblastoma and patients with Hodgkin's lymphoma, and phase II part patients with relapsed or refractory glioblastoma.

A separate Japanese single agent dose escalation was performed in order to ensure that the safety and pharmacokinetic profiles of BLZ945 single agent were adequately characterized in Japanese patients. The Japanese dose escalation for BLZ945 single agent run separately from the ongoing global dose escalation. No Japanese patients were enrolled in phase II part according to protocol. The enrollment of the Japanese cohort was halted per investigator letter, dated 18-Jun-2021.

ELIGIBILITY:
Inclusion Criteria:

1. Phase I: Patients with advanced/metastatic solid tumors including relapsed or refractory (r/r) glioblastoma and r/r lymphoma, with measurable or unmeasurable disease as determined by the respective response evaluation criteria.
2. Phase I: Patients with a site of disease amenable to biopsy, and willing to undergo a new tumor biopsy at screening, and during treatment.
3. Phase II: Patients with advanced/metastatic/recurrent isocitrate dehydrogenase (IDH) wild-type glioblastoma, with at least one measurable lesion as determined by RANO

Exclusion Criteria:

1. History of severe hypersensitivity reactions to monoclonal antibodies.
2. Impaired cardiac function or clinically significant cardiac disease.
3. Active autoimmune disease or a documented history of autoimmune disease.
4. Systemic steroid therapy or any immunosuppressive therapy
5. Use of any vaccines against infectious diseases within 4 weeks of initiation of study treatment.
6. Patient receiving treatment with medications that either strong inducers or inhibitors of CYP2C8 or CYP3A4/5, or patients receiving medication that prohibits proton pump inhibitors and that cannot be discontinued at least 1 week prior to start of treatment and for the duration of the study.
7. Presence of symptomatic central nervous system (CNS) metastases, or CNS metastases that require local CNS-directed therapy (such as radiotherapy or surgery), or increasing doses of corticosteroids within the prior 2 weeks before start of study treatment (not applicable for glioblastoma).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- United States (4):
  - Dana Farber Cancer Institute Dana Farber Cancer Institute, Boston, Massachusetts
  - Sarah Cannon Research Institute Sarah Cannon Research, Nashville, Tennessee
  - UT M.D Anderson Cancer Center, Houston, Texas
  - Mays Cancer Ctr Uthsa Mdacc, San Antonio, Texas
- Novartis Investigative Site, Tel Aviv, Israel
- Novartis Investigative Site, Rozzano, MI, Italy
- Japan (2):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Koto Ku, Tokyo
- Novartis Investigative Site, Singapore, Singapore
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Zurich, Switzerland
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 14 investigative sites in 8 countries.
Pre-assignment Details: The screening period began once patients had signed the study informed consent. Screening evaluations were performed within 28 days prior to the first dose of study medication. After screening, the treatment period started on Cycle 1 Day 1.
Groups:
- Phase I: BLZ945 150 mg 7d on/7d Off QD: BLZ945 150 mg once per day administered for 7 days and suspended for 7 days
- Phase I: BLZ945 300 mg 7d on/7d Off QD: BLZ945 300 mg once per day administered for 7 days and suspended for 7 days
- Phase I: BLZ945 300 mg Q1W QD: BLZ945 300 mg once per day once weekly
- Phase I: BLZ945 450 mg Q1W QD: BLZ945 450 mg once per day once weekly
- Phase I: BLZ945 600 mg Q1W QD: BLZ945 600 mg once per day once weekly
- Phase I: BLZ945 1000 mg Q1W QD: BLZ945 1000 mg once per day once weekly
- Phase I: BLZ945 1600 mg Q1W QD: BLZ945 1600 mg once per day once weekly
- Phase I: BLZ945 300 mg 4d on/10d Off QD: BLZ945 300 mg once per day administered for 4 days and suspended for 10 days
- Phase I: BLZ945 600 mg 4d on/10d Off QD: BLZ945 600 mg once per day administered for 4 days and suspended for 10 days
- Phase I: BLZ945 800 mg 4d on/10d Off QD: BLZ945 800 mg once per day administered for 4 days and suspended for 10 days
- Phase I: BLZ945 1200 mg 4d on/10d Off QD; Phase II: BLZ945 1200 mg 4d on/10d Off QD: BLZ945 1200 mg once per day administered for 4 days and suspended for 10 days
- Phase I: BLZ945 300 mg Q1W BID: BLZ945 300 mg twice per day once weekly
- Phase I: BLZ945 600 mg Q1W BID: BLZ945 600 mg twice per day once weekly
- Phase I: BLZ945 600 mg 4d on/10d Off BID: BLZ945 600 mg twice per day administered for 4 days and suspended for 10 days
- Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W: BLZ945 150 mg once per day once weekly in combination with PDR001 400 mg every 4 weeks
- Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W: BLZ945 300 mg once per day once weekly in combination with PDR001 400 mg every 4 weeks
- Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W: BLZ945 600 mg once per day once weekly in combination with PDR001 400 mg every 4 weeks
- Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W: BLZ945 1000 mg once per day once weekly in combination with PDR001 400 mg every 4 weeks
- Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W: BLZ945 1400 mg once per day once weekly in combination with PDR001 400 mg every 4 weeks
- Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W: BLZ945 300 mg once per day administered for 4 days and suspended for 10 days in combination with PDR001 400 mg every 4 weeks
- Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W: BLZ945 450 mg once per day administered for 4 days and suspended for 10 days in combination with PDR001 400 mg every 4 weeks
- Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W; Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W: BLZ945 700 mg once per day administered for 4 days and suspended for 10 days in combination with PDR001 400 mg every 4 weeks
- Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W: BLZ945 1200 mg once per day administered for 4 days and suspended for 10 days in combination with PDR001 400 mg every 4 weeks
- Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W: BLZ945 600 mg twice per day once weekly in combination with PDR001 400 mg every 4 weeks
- Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W: BLZ945 800 mg twice per day once weekly in combination with PDR001 400 mg every 4 weeks
Period: Overall Study
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W | Phase II: BLZ945 1200 mg 4d on/10d Off QD | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W
Started (The Full Analysis Set (FAS) comprises all patients who received at least one dose of study treatment. Patients were analyzed according to the planned treatment.) | 5 | 7 | 5 | 6 | 3 | 5 | 6 | 8 | 9 | 5 | 10 | 0 | 5 | 6 | 4 | 5 | 9 | 5 | 6 | 5 | 11 | 9 | 4 | 6 | 5 | 22 | 21
Safety Set (The Safety Set includes all patients who received at least one dose of BLZ945 or PDR001. Patients were analyzed according to the study treatment (regimen) they actually received.) | 5 | 7 | 5 | 6 | 3 | 5 | 6 | 8 | 9 | 5 | 10 | 1 | 4 | 6 | 4 | 5 | 9 | 5 | 6 | 5 | 11 | 9 | 4 | 6 | 5 | 22 | 21
Japanese Cohort | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 7 | 5 | 6 | 3 | 5 | 6 | 8 | 9 | 5 | 10 | 0 | 5 | 6 | 4 | 5 | 9 | 5 | 6 | 5 | 11 | 9 | 4 | 6 | 5 | 22 | 21
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 1 | 3 | 0 | 0 | 1 | 1 | 3 | 5
Not completed — Death | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3
Not completed — Progressive disease | 4 | 6 | 3 | 3 | 3 | 5 | 4 | 6 | 8 | 4 | 9 | 0 | 3 | 4 | 2 | 4 | 5 | 3 | 4 | 4 | 7 | 6 | 3 | 3 | 3 | 16 | 10
Not completed — Subject/guardian decision | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W | Phase II: BLZ945 1200 mg 4d on/10d Off QD | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Total
Number analyzed (Participants) | 5 | 7 | 5 | 6 | 3 | 5 | 6 | 8 | 9 | 5 | 10 | 5 | 6 | 4 | 5 | 9 | 5 | 6 | 5 | 11 | 9 | 4 | 6 | 5 | 22 | 21 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (9.42) | 55.0 (17.68) | 59.2 (13.33) | 55.3 (9.40) | 59.0 (3.61) | 55.4 (18.85) | 60.7 (14.24) | 55.5 (15.11) | 54.6 (17.48) | 57.6 (6.95) | 63.0 (8.94) | 52.8 (15.64) | 57.0 (16.80) | 53.5 (18.77) | 59.6 (3.21) | 46.7 (9.11) | 58.2 (13.52) | 50.7 (16.68) | 49.8 (19.77) | 58.9 (13.26) | 50.6 (15.42) | 46.3 (15.59) | 67.2 (9.37) | 53.2 (13.31) | 56.8 (12.64) | 55.0 (8.79) | 55.7 (13.12)
Age, Customized [Count of Participants; unit: Participants]
  18 - < 65 years | 5 | 5 | 4 | 5 | 3 | 3 | 3 | 6 | 6 | 4 | 5 | 4 | 3 | 2 | 5 | 9 | 3 | 5 | 3 | 6 | 7 | 3 | 1 | 4 | 15 | 19 | 138
  65 - < 85 years | 0 | 2 | 1 | 1 | 0 | 2 | 3 | 2 | 3 | 1 | 5 | 1 | 3 | 2 | 0 | 0 | 2 | 1 | 2 | 5 | 2 | 1 | 5 | 1 | 7 | 2 | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 3 | 0 | 4 | 3 | 4 | 5 | 3 | 5 | 0 | 2 | 3 | 2 | 4 | 1 | 2 | 2 | 4 | 2 | 2 | 3 | 3 | 8 | 6 | 79
  Male | 3 | 4 | 2 | 3 | 3 | 1 | 3 | 4 | 4 | 2 | 5 | 5 | 4 | 1 | 3 | 5 | 4 | 4 | 3 | 7 | 7 | 2 | 3 | 2 | 14 | 15 | 113
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 5 | 1 | 1 | 2 | 0 | 1 | 3 | 6 | 1 | 2 | 0 | 2 | 1 | 1 | 4 | 0 | 3 | 2 | 3 | 2 | 2 | 3 | 1 | 1 | 1 | 49
  Black or African American | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 7
  White | 4 | 2 | 4 | 2 | 1 | 5 | 5 | 5 | 3 | 4 | 7 | 4 | 4 | 3 | 4 | 4 | 5 | 3 | 3 | 6 | 6 | 2 | 3 | 4 | 20 | 20 | 133
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) During the On-treatment Period
Description: Number of participants with AEs (any AE regardless of seriousness) and SAEs, including changes from baseline in vital signs, electrocardiograms and laboratory results qualifying and reported as AEs.
  The on-treatment period is defined from the day of first administration of study treatment up to 30 days after the date of its last administration.
Time Frame: From first dose of study medication up to 30 days after last dose, with a maximum duration of 3.1 years for BLZ945 single agent and 4.1 years for BLZ945 in combination with PDR001
Population: All patients from Phase I who received at least one dose of BLZ945 or PDR001. Patients were analyzed according to the study treatment (regimen) they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 5 | 7 | 5 | 6 | 3 | 5 | 6 | 8 | 9 | 5 | 10 | 1 | 4 | 6 | 4 | 5 | 9 | 5 | 6 | 5 | 11 | 9 | 4 | 6 | 5
Participants
  AEs | 5 | 7 | 5 | 6 | 3 | 5 | 6 | 8 | 9 | 5 | 10 | 1 | 4 | 6 | 4 | 5 | 9 | 5 | 6 | 5 | 11 | 9 | 4 | 6 | 5
  Treatment-related AEs | 3 | 7 | 5 | 4 | 3 | 5 | 5 | 6 | 8 | 4 | 7 | 0 | 4 | 6 | 2 | 4 | 7 | 5 | 4 | 4 | 8 | 4 | 4 | 5 | 4
  SAEs | 3 | 1 | 3 | 2 | 0 | 3 | 3 | 4 | 3 | 3 | 5 | 0 | 3 | 5 | 1 | 1 | 5 | 4 | 3 | 1 | 5 | 7 | 4 | 2 | 1
  Treatment-related SAEs | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 1
  Fatal SAEs | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0

2. Primary Outcome: Phase I: Number of Participants With Dose Reductions and Dose Interruptions of BLZ945
Description: Number of participants with at least one dose reduction of BLZ945 and number of participants with at least one dose interruption of BLZ945.
Time Frame: From first dose of study medication up to last dose, with a maximum duration of 3 years for BLZ945 single agent and 4 years for BLZ945 in combination with PDR001
Population: All patients from Phase I who received at least one dose of BLZ945. Patients were analyzed according to the study treatment (regimen) they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 5 | 7 | 5 | 6 | 3 | 5 | 6 | 8 | 9 | 5 | 10 | 1 | 4 | 6 | 4 | 5 | 9 | 5 | 6 | 5 | 11 | 9 | 4 | 6 | 5
Participants
  At least one dose reduction | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 2
  At least one dose interruption | 4 | 2 | 2 | 3 | 1 | 3 | 1 | 2 | 0 | 2 | 5 | 0 | 1 | 1 | 0 | 1 | 4 | 2 | 3 | 1 | 4 | 6 | 2 | 2 | 1

3. Primary Outcome: Phase I: Number of Participants With Dose Reductions and Dose Interruptions of PDR001
Description: Number of participants with at least one dose reduction of PDR001 and number of participants with at least one dose interruption of PDR001. Dose reductions were not permitted for PDR001.
Time Frame: From first dose of study medication up to last dose, with a maximum duration of 4 years
Population: All patients from Phase I who received at least one dose of PDR001. Patients were analyzed according to the study treatment (regimen) they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 4 | 5 | 9 | 5 | 6 | 5 | 11 | 9 | 4 | 6 | 5
Participants
  At least one dose reduction | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  At least one dose interruption | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 0 | 1 | 1

4. Primary Outcome: Phase I: Dose Intensity of BLZ945
Description: Dose intensity of BLZ945 was calculated as cumulative actual dose in milligrams divided by the number of dose days scheduled per protocol during the treatment period. The denominator was calculated considering that patients received doses 7 days out of every 14 in the 7 days on/7 days off regimen, 4 days out of every 14 in the 4 days on/10 days off regimen and 1 day out of every 7 in the Q1W regimen.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 5 | 7 | 5 | 6 | 3 | 5 | 6 | 8 | 9 | 5 | 10 | 1 | 4 | 6 | 4 | 5 | 9 | 5 | 6 | 5 | 11 | 9 | 4 | 6 | 5
mg/day | 141.4 (5.16) | 250.1 (39.30) | 281.8 (52.50) | 399.2 (63.71) | 525.0 (129.90) | 959.5 (132.40) | 1570.9 (153.93) | 277.8 (25.70) | 578.8 (27.27) | 705.1 (98.99) | 1055.0 (103.62) | 600.0 | 1063.1 (321.62) | 1105.5 (71.77) | 160.0 (14.14) | 293.5 (14.50) | 566.3 (51.79) | 945.7 (87.13) | 1259.0 (209.04) | 286.0 (18.49) | 416.1 (32.30) | 606.9 (56.03) | 862.0 (243.73) | 1125.1 (224.13) | 1448.0 (386.16)

5. Primary Outcome: Phase I: Dose Intensity of PDR001
Description: Dose intensity of PDR001 was calculated as cumulative actual dose in milligrams divided by the number of dose days scheduled per protocol during the treatment period. The denominator was calculated considering that patients received doses 1 day out of every 28 in the Q4W regimen.
Time Frame: From first dose of study medication up to last dose, with a maximum duration of 4 years
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 4 | 5 | 9 | 5 | 6 | 5 | 11 | 9 | 4 | 6 | 5
mg/day | 533.3 (188.56) | 400.0 (0.00) | 400.0 (0.00) | 426.7 (59.63) | 433.3 (81.65) | 420.0 (44.72) | 390.5 (31.46) | 393.1 (14.05) | 400.0 (0.00) | 466.7 (163.30) | 453.3 (202.21)

6. Primary Outcome: Phase I: Number of Participants With Dose-Limiting Toxicities (DLTs) (Non-Japanese Cohort)
Description: A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value of Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 3 assessed as unrelated to disease, disease progression, inter-current illness or concomitant medications, which occurs within the first 28 days of treatment with BLZ945 as single agent or in combination with PDR001 during the dose escalation part of the study. Other clinically significant toxicities may be considered to be DLTs, even if not CTCAE grade 3 or higher.
Time Frame: 28 days
Population: Non-Japanese patients in Phase I who either met the minimum exposure criterion defined in the protocol and had sufficient safety evaluations, or had experienced a DLT during Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 5 | 7 | 5 | 6 | 3 | 5 | 6 | 5 | 4 | 4 | 9 | 0 | 4 | 6 | 4 | 5 | 9 | 5 | 6 | 5 | 11 | 8 | 3 | 6 | 4
Participants | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 |  | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 2

7. Primary Outcome: Phase I: Number of Participants With Dose-Limiting Toxicities (DLTs) (Japanese Cohort)
Description: as for outcome 6
Time Frame: 28 days
Population: Japanese patients in Phase I who either met the minimum exposure criterion defined in the protocol and had sufficient safety evaluations, or had experienced a DLT during Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 0 | 0 | 0 | 0 | 0
Participants |  |  |  |  |  |  |  | 0 | 1 |  |  |  |  |

8. Primary Outcome: Phase II: Progression-Free Survival Rate at 6 Months (PFS6) Per RANO Criteria for Glioblastoma
Description: PFS rate represents the percentage of participants without a first documented progression or death due to any cause after the start of study treatment. Tumor response was based on local investigator assessment per Response Assessment in Neuro Oncology (RANO) criteria.
  PFS was analyzed using Kaplan-Meier estimates.
Time Frame: 6 months
Population: All patients from Phase II who received at least one dose of BLZ945 or PDR001. Patients were analyzed according to the planned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: BLZ945 1200 mg 4d on/10d Off QD | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W
Number analyzed (Participants) | 22 | 21
percentage of participants | 15.2 [3.8 to 33.9] | 22.2 [7.1 to 42.6]

9. Secondary Outcome: Phase I: Progression-Free Survival (PFS) Per RECIST v1.1
Description: PFS is defined as the time from the date of start of treatment to the date of the first documented progression or death due to any cause. If a patient did not have an event, PFS was censored at the date of the last adequate tumor assessment. Tumor response was based on local investigator assessment per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.
  PFS was analyzed using Kaplan-Meier estimates.
Time Frame: From start of treatment until first documented progression or death due to any cause, assessed up to 3.1 years for BLZ945 single agent and 4.4 years for BLZ945 in combination with PDR001
Population: All patients from Phase I with solid tumors (excluding glioblastoma and lymphoma) who received at least one dose of BLZ945 or PDR001. Patients were analyzed according to the planned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 5 | 7 | 5 | 6 | 3 | 5 | 5 | 8 | 8 | 5 | 7 | 0 | 1 | 3 | 4 | 5 | 7 | 5 | 5 | 4 | 6 | 4 | 3 | 6 | 3
months | NA [1.6 to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [1.7 to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [1.7 to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | 1.9 [1.8 to NA] — Not estimable due to insufficient number of participants with events. | NA [1.8 to NA] — Not estimable due to insufficient number of participants with events. |  | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | 7.9 [1.9 to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [1.9 to NA] — Not estimable due to insufficient number of participants with events. | 3.5 [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [1.1 to NA] — Not estimable due to insufficient number of participants with events. | NA [1.8 to NA] — Not estimable due to insufficient number of participants with events. | 40.1 [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [0.0 to NA] — Not estimable due to insufficient number of participants with events. | NA [0.0 to NA] — Not estimable due to insufficient number of participants with events. | NA [1.8 to NA] — Not estimable due to insufficient number of participants with events.

10. Secondary Outcome: Phase I: Progression-Free Survival (PFS) Per irRC
Description: PFS is defined as the time from the date of start of treatment to the date of the first documented progression or death due to any cause. If a patient did not have an event, PFS was censored at the date of the last adequate tumor assessment. Tumor response was based on local investigator assessment per immune-related Response Criteria (irRC).
  PFS was analyzed using Kaplan-Meier estimates.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 5 | 7 | 5 | 6 | 3 | 5 | 5 | 8 | 8 | 5 | 7 | 0 | 1 | 3 | 4 | 5 | 7 | 5 | 5 | 4 | 6 | 4 | 3 | 6 | 3
months | NA [1.6 to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [1.7 to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [1.7 to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | 1.9 [1.8 to NA] — Not estimable due to insufficient number of participants with events. | NA [1.8 to NA] — Not estimable due to insufficient number of participants with events. |  | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | 7.9 [1.9 to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [1.9 to NA] — Not estimable due to insufficient number of participants with events. | 3.5 [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [1.1 to NA] — Not estimable due to insufficient number of participants with events. | NA [1.8 to NA] — Not estimable due to insufficient number of participants with events. | 40.1 [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [0.0 to NA] — Not estimable due to insufficient number of participants with events. | 2.6 [0.0 to NA] — Not estimable due to insufficient number of participants with events. | NA [1.8 to NA] — Not estimable due to insufficient number of participants with events.

11. Secondary Outcome: Phase I: Progression-Free Survival (PFS) Per RANO
Description: PFS is defined as the time from the date of start of treatment to the date of the first documented progression or death due to any cause. If a patient did not have an event, PFS was censored at the date of the last adequate tumor assessment. Tumor response was based on local investigator assessment per response assessment in neuro-oncology (RANO) criteria.
  PFS was analyzed using Kaplan-Meier estimates.
Time Frame: as for outcome 9
Population: All patients from Phase I with glioblastoma who received at least one dose of BLZ945 or PDR001. Patients were analyzed according to the planned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 4 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 3 | 1 | 0 | 2
months |  |  |  |  |  |  | 1.9 [NA to NA] — Not estimable due to insufficient number of participants with events. |  | 0.2 [NA to NA] — Not estimable due to insufficient number of participants with events. |  | 1.9 [1.3 to NA] — Not estimable due to insufficient number of participants with events. |  | 2.8 [0.2 to NA] — Not estimable due to insufficient number of participants with events. | 1.9 [1.9 to NA] — Not estimable due to insufficient number of participants with events. |  |  |  |  | 1.9 [NA to NA] — Not estimable due to insufficient number of participants with events. | 3.6 [NA to NA] — Not estimable due to insufficient number of participants with events. | 1.9 [1.4 to NA] — Not estimable due to insufficient number of participants with events. | 0.7 [0.5 to NA] — Not estimable due to insufficient number of participants with events. | 0.8 [NA to NA] — Not estimable due to insufficient number of participants with events. |  | 1.1 [0.3 to NA] — Not estimable due to insufficient number of participants with events.

12. Secondary Outcome: Phase I and II: Progression-Free Survival (PFS) Per iRANO
Description: PFS is defined as the time from the date of start of treatment to the date of the first documented progression or death due to any cause. If a patient did not have an event, PFS was censored at the date of the last adequate tumor assessment. Tumor response was based on local investigator assessment per immune response assessment in neuro-oncology (iRANO) criteria.
  PFS was analyzed using Kaplan-Meier estimates.
Time Frame: as for outcome 9
Population: All patients with glioblastoma who received at least one dose of BLZ945 or PDR001. Patients were analyzed according to the planned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W | Phase II: BLZ945 1200 mg 4d on/10d Off QD | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 4 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 3 | 1 | 0 | 2 | 22 | 21
months |  |  |  |  |  |  | NA [NA to NA] — Not estimable due to insufficient number of participants with events. |  | NA [NA to NA] — Not estimable due to insufficient number of participants with events. |  | NA [NA to NA] — Not estimable due to insufficient number of participants with events. |  | NA [1.6 to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. |  |  |  |  | 2.2 [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | 12.0 [3.6 to NA] — Not estimable due to insufficient number of participants with events. | 1.2 [0.5 to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. |  | 3.2 [NA to NA] — Not estimable due to insufficient number of participants with events. | 6.7 [1.1 to NA] — Not estimable due to insufficient number of participants with events. | 3.0 [1.3 to NA] — Not estimable due to insufficient number of participants with events.

13. Secondary Outcome: Phase I: Progression-Free Survival (PFS) Per Guidelines for Efficacy Evaluation in Lymphoma Studies
Description: PFS is defined as the time from the date of start of treatment to the date of the first documented progression or death due to any cause. If a patient did not have an event, PFS was censored at the date of the last adequate tumor assessment. Tumor response was based on local investigator assessment per guidelines for efficacy evaluation in lymphoma studies.
  PFS was analyzed using Kaplan-Meier estimates.
Time Frame: as for outcome 9
Population: All patients from Phase I with lymphoma who received at least one dose of BLZ945 or PDR001. Patients were analyzed according to the planned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
months |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | NA [NA to NA] — Not estimable due to insufficient number of participants with events. |  |  |  |  | 2.2 [1.5 to NA] — Not estimable due to insufficient number of participants with events. |  |  |

14. Secondary Outcome: Phase I: Best Overall Response (BOR) With Confirmation Per RECIST v1.1
Description: BOR is defined as the best response recorded from the start of the study treatment until disease progression/recurrence, based on local investigator assessment per RECIST v1.1. However, any assessments taken more than 30 days after the last dose of study therapy were not included in the best overall response derivation.
  Complete Response (CR) and Partial response (PR) had to be confirmed by a new assessment after at least 4 weeks.
Time Frame: From start of treatment until disease progression, assessed up to 3.1 years for BLZ945 single agent and 4.1 years for BLZ945 in combination with PDR001
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 5 | 7 | 5 | 6 | 3 | 5 | 5 | 8 | 8 | 5 | 7 | 0 | 1 | 3 | 4 | 5 | 7 | 5 | 5 | 4 | 6 | 4 | 3 | 6 | 3
Participants
  Complete Response (CR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Stable Disease (SD) | 3 | 1 | 1 | 4 | 0 | 2 | 0 | 4 | 3 | 2 | 2 |  | 0 | 1 | 3 | 2 | 3 | 1 | 2 | 2 | 2 | 4 | 0 | 1 | 1
  Progressive Disease (PD) | 1 | 6 | 4 | 0 | 3 | 3 | 3 | 4 | 4 | 3 | 4 |  | 1 | 2 | 1 | 3 | 3 | 3 | 3 | 1 | 3 | 0 | 2 | 4 | 2
  Unknown | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 1 |  | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0
  Non-CR/Non-PD (NCRNPD) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Phase I: Best Overall Response (BOR) With Confirmation Per irRC
Description: BOR is defined as the best response recorded from the start of the study treatment until disease progression/recurrence, based on local investigator assessment per irRC. However, any assessments taken more than 30 days after the last dose of study therapy were not included in the best overall response derivation.
  Complete Response (CR) and Partial response (PR) had to be confirmed by a new assessment after at least 4 weeks. Additionally, for irRC, progressive disease had to be confirmed.
Time Frame: as for outcome 14
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 5 | 7 | 5 | 6 | 3 | 5 | 5 | 8 | 8 | 5 | 7 | 0 | 1 | 3 | 4 | 5 | 7 | 5 | 5 | 4 | 6 | 4 | 3 | 6 | 3
Participants
  Complete Response (irCR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response (irPR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Stable Disease (irSD) | 3 | 1 | 1 | 4 | 0 | 2 | 0 | 4 | 3 | 2 | 2 |  | 0 | 1 | 3 | 2 | 3 | 1 | 2 | 2 | 2 | 4 | 0 | 2 | 1
  Progressive Disease (irPD) | 1 | 6 | 4 | 0 | 3 | 3 | 3 | 4 | 4 | 3 | 4 |  | 1 | 2 | 1 | 3 | 3 | 3 | 3 | 1 | 3 | 0 | 2 | 3 | 2
  Unknown | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 1 |  | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0

16. Secondary Outcome: Phase I and II: Best Overall Response (BOR) (Sustained) Per RANO
Description: BOR is defined as the best response recorded from the start of the study treatment until disease progression (taking as reference for progressive disease the smallest measurements recorded since the treatment started), based on local investigator assessment per RANO criteria. However, any assessments taken more than 30 days after the last dose of study therapy were not included in the best overall response derivation.
  If a response recorded at one scheduled magnetic resonance imaging (MRI) did not persist at the next regular scheduled MRI, the response was recorded based on the prior scan, but was designated as a non-sustained response. If the response was sustained, i.e. still present on the subsequent MRI, it was recorded as a sustained response, lasting until the time of tumor progression. CR and PR had to be confirmed by repeat assessments performed not less than 4 weeks after the criteria for response were first met.
Time Frame: From start of treatment until disease progression, assessed up to 4.1 years in Phase I and 1.4 years in Phase II
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W | Phase II: BLZ945 1200 mg 4d on/10d Off QD | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 4 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 3 | 1 | 0 | 2 | 22 | 21
Participants
  Complete Response (CR) |  |  |  |  |  |  | 0 |  | 0 |  | 0 |  | 0 | 0 |  |  |  |  | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Partial Response (PR) |  |  |  |  |  |  | 0 |  | 0 |  | 1 |  | 0 | 0 |  |  |  |  | 0 | 0 | 0 | 0 | 0 |  | 0 | 3 | 0
  Stable Disease (SD) |  |  |  |  |  |  | 0 |  | 0 |  | 0 |  | 2 | 1 |  |  |  |  | 0 | 1 | 2 | 0 | 0 |  | 0 | 3 | 5
  Progressive Disease (PD) as per tumor assessment |  |  |  |  |  |  | 1 |  | 0 |  | 2 |  | 0 | 1 |  |  |  |  | 1 | 0 | 3 | 2 | 1 |  | 1 | 10 | 11
  Progressive Disease (PD) as per clinical assessment |  |  |  |  |  |  | 0 |  | 1 |  | 0 |  | 1 | 1 |  |  |  |  | 0 | 0 | 0 | 0 | 0 |  | 1 | 4 | 1
  Unknown |  |  |  |  |  |  | 0 |  | 0 |  | 0 |  | 1 | 0 |  |  |  |  | 0 | 0 | 0 | 1 | 0 |  | 0 | 2 | 4

17. Secondary Outcome: Phase I and II: Best Overall Response (BOR) (Sustained) Per iRANO
Description: BOR is defined as the best response recorded from the start of the study treatment until disease progression (taking as reference for progressive disease the smallest measurements recorded since the treatment started), based on local investigator assessment per iRANO. However, any assessments taken more than 30 days after the last dose of study therapy were not included in the best overall response derivation.
  If a response recorded at one scheduled magnetic resonance imaging (MRI) did not persist at the next regular scheduled MRI, the response was recorded based on the prior scan, but was designated as a non-sustained response. If the response was sustained, i.e. still present on the subsequent MRI, it was recorded as a sustained response, lasting until the time of tumor progression. CR and PR had to be confirmed by repeat assessments performed not less than 4 weeks after the criteria for response were first met. Additionally, for iRANO, progressive disease had to be confirmed.
Time Frame: From start of treatment until disease progression, assessed up to 4.1 years in Phase I and 1.4 years in Phase II
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W | Phase II: BLZ945 1200 mg 4d on/10d Off QD | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 4 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 3 | 1 | 0 | 2 | 22 | 21
Participants
  Complete Response (CR) |  |  |  |  |  |  | 0 |  | 0 |  | 0 |  | 0 | 0 |  |  |  |  | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Partial Response (PR) |  |  |  |  |  |  | 0 |  | 0 |  | 1 |  | 0 | 0 |  |  |  |  | 0 | 1 | 0 | 0 | 0 |  | 0 | 3 | 0
  Stable Disease (SD) |  |  |  |  |  |  | 0 |  | 0 |  | 0 |  | 2 | 1 |  |  |  |  | 0 | 0 | 2 | 0 | 0 |  | 0 | 3 | 5
  Progressive Disease (PD) as per tumor assessment |  |  |  |  |  |  | 0 |  | 0 |  | 0 |  | 0 | 0 |  |  |  |  | 0 | 0 | 0 | 1 | 0 |  | 0 | 1 | 0
  Progressive Disease (PD) as per clinical assessment |  |  |  |  |  |  | 0 |  | 0 |  | 0 |  | 0 | 0 |  |  |  |  | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Unknown |  |  |  |  |  |  | 1 |  | 1 |  | 2 |  | 2 | 2 |  |  |  |  | 1 | 0 | 3 | 2 | 1 |  | 2 | 15 | 16

18. Secondary Outcome: Phase I: Best Overall Response (BOR) Per Guidelines for Efficacy Evaluation in Lymphoma Studies
Description: BOR is defined as the best response recorded from the start of the study treatment until disease progression/recurrence, based on local investigator assessment per guidelines for efficacy evaluation in lymphoma studies. However, any assessments taken more than 30 days after the last dose of study therapy were not included in the best overall response derivation.
Time Frame: as for outcome 14
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Participants
  Complete Response (CR) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  |  |  |  | 0 |  |  |
  Partial response (PR) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  |  |  |  | 1 |  |  |
  Stable disease (SD) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  |  |  |  | 0 |  |  |
  Progressive Disease (PD) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  |  |  |  | 1 |  |  |
  Unknown |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 2 |  |  |  |  | 0 |  |  |

19. Secondary Outcome: Phase I: Overall Response Rate (ORR) Per RECIST v1.1
Description: ORR is the percentage of patients with a best overall response of complete response (CR) or partial response (PR), based on local investigator assessment per RECIST v1.1.
Time Frame: Up to 3.1 years for BLZ945 single agent and 4.1 years for BLZ945 in combination with PDR001
Population: as for outcome 9
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 5 | 7 | 5 | 6 | 3 | 5 | 5 | 8 | 8 | 5 | 7 | 0 | 1 | 3 | 4 | 5 | 7 | 5 | 5 | 4 | 6 | 4 | 3 | 6 | 3
percentage of participants | 0 [0.0 to 45.1] | 0 [0.0 to 34.8] | 0 [0.0 to 45.1] | 0 [0.0 to 39.3] | 0 [0.0 to 63.2] | 0 [0.0 to 45.1] | 0 [0.0 to 45.1] | 0 [0.0 to 31.2] | 0 [0.0 to 31.2] | 0 [0.0 to 45.1] | 0 [0.0 to 34.8] |  | 0 [0.0 to 95.0] | 0 [0.0 to 63.2] | 0 [0.0 to 52.7] | 0 [0.0 to 45.1] | 14.3 [0.7 to 52.1] | 0 [0.0 to 45.1] | 0 [0.0 to 45.1] | 0 [0.0 to 52.7] | 0 [0.0 to 39.3] | 0 [0.0 to 52.7] | 0 [0.0 to 63.2] | 0 [0.0 to 39.3] | 0 [0.0 to 63.2]

20. Secondary Outcome: Phase I: Overall Response Rate (ORR) Per irRC
Description: ORR is the percentage of patients with a best overall response of complete response (irCR) or partial response (irPR), based on local investigator assessment per irRC.
Time Frame: Up to 3.1 years for BLZ945 single agent and 4.1 years for BLZ945 in combination with PDR001
Population: as for outcome 9
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 5 | 7 | 5 | 6 | 3 | 5 | 5 | 8 | 8 | 5 | 7 | 0 | 1 | 3 | 4 | 5 | 7 | 5 | 5 | 4 | 6 | 4 | 3 | 6 | 3
percentage of participants | 0 [0.0 to 45.1] | 0 [0.0 to 34.8] | 0 [0.0 to 45.1] | 0 [0.0 to 39.3] | 0 [0.0 to 63.2] | 0 [0.0 to 45.1] | 0 [0.0 to 45.1] | 0 [0.0 to 31.2] | 0 [0.0 to 31.2] | 0 [0.0 to 45.1] | 0 [0.0 to 34.8] |  | 0 [0.0 to 95.0] | 0 [0.0 to 63.2] | 0 [0.0 to 52.7] | 0 [0.0 to 45.1] | 14.3 [0.7 to 52.1] | 0 [0.0 to 45.1] | 0 [0.0 to 45.1] | 0 [0.0 to 52.7] | 0 [0.0 to 39.3] | 0 [0.0 to 52.7] | 0 [0.0 to 63.2] | 0 [0.0 to 39.3] | 0 [0.0 to 63.2]

21. Secondary Outcome: Phase I: Overall Response Rate (ORR) Per Guidelines for Efficacy Evaluation in Lymphoma Studies
Description: ORR is the percentage of patients with a best overall response of complete response (CR) or partial response (PR), based on local investigator assessment per guidelines for efficacy evaluation in lymphoma studies.
Time Frame: Up to 3.1 years for BLZ945 single agent and 4.1 years for BLZ945 in combination with PDR001
Population: as for outcome 13
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
percentage of participants |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0 [0.0 to 77.6] |  |  |  |  | 50.0 [2.5 to 97.5] |  |  |

22. Secondary Outcome: Phase I: Disease Control Rate (DCR) Per RECIST v1.1
Description: DCR is the percentage of patients with a best overall response of complete response (CR), partial response (PR) or stable disease (SD), based on local investigator assessment per RECIST v1.1.
Time Frame: Up to 3.1 years for BLZ945 single agent and 4.1 years for BLZ945 in combination with PDR001
Population: as for outcome 9
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 5 | 7 | 5 | 6 | 3 | 5 | 5 | 8 | 8 | 5 | 7 | 0 | 1 | 3 | 4 | 5 | 7 | 5 | 5 | 4 | 6 | 4 | 3 | 6 | 3
percentage of participants | 60.0 [18.9 to 92.4] | 14.3 [0.7 to 52.1] | 20.0 [1.0 to 65.7] | 66.7 [27.1 to 93.7] | 0 [0.0 to 63.2] | 40.0 [7.6 to 81.1] | 0 [0.0 to 45.1] | 50.0 [19.3 to 80.7] | 37.5 [11.1 to 71.1] | 40.0 [7.6 to 81.1] | 28.6 [5.3 to 65.9] |  | 0 [0.0 to 95.0] | 33.3 [1.7 to 86.5] | 75.0 [24.9 to 98.7] | 40.0 [7.6 to 81.1] | 57.1 [22.5 to 87.1] | 20.0 [1.0 to 65.7] | 40.0 [7.6 to 81.1] | 50.0 [9.8 to 90.2] | 33.3 [6.3 to 72.9] | 100 [47.3 to 100.0] | 0 [0.0 to 63.2] | 16.7 [0.9 to 58.2] | 33.3 [1.7 to 86.5]

23. Secondary Outcome: Phase I: Disease Control Rate (DCR) Per irRC
Description: DCR is the percentage of patients with a best overall response of complete response (irCR), partial response (irPR) or stable disease (irSD), based on local investigator assessment per irRC.
Time Frame: Up to 3.1 years for BLZ945 single agent and 4.1 years for BLZ945 in combination with PDR001
Population: as for outcome 9
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 5 | 7 | 5 | 6 | 3 | 5 | 5 | 8 | 8 | 5 | 7 | 0 | 1 | 3 | 4 | 5 | 7 | 5 | 5 | 4 | 6 | 4 | 3 | 6 | 3
percentage of participants | 60.0 [18.9 to 92.4] | 14.3 [0.7 to 52.1] | 20.0 [1.0 to 65.7] | 66.7 [27.1 to 93.7] | 0 [0.0 to 63.2] | 40.0 [7.6 to 81.1] | 0 [0.0 to 45.1] | 50.0 [19.3 to 80.7] | 37.5 [11.1 to 71.1] | 40.0 [7.6 to 81.1] | 28.6 [5.3 to 65.9] |  | 0 [0.0 to 95.0] | 33.3 [1.7 to 86.5] | 75.0 [24.9 to 98.7] | 40.0 [7.6 to 81.1] | 57.1 [22.5 to 87.1] | 20.0 [1.0 to 65.7] | 40.0 [7.6 to 81.1] | 50.0 [9.8 to 90.2] | 33.3 [6.3 to 72.9] | 100 [47.3 to 100] | 0 [0.0 to 63.2] | 33.3 [6.3 to 72.9] | 33.3 [1.7 to 86.5]

24. Secondary Outcome: Phase I and II: Disease Control Rate (DCR) Per RANO
Description: DCR is the percentage of patients with a best overall response of complete response (CR), partial response (PR) or stable disease (SD), based on local investigator assessment per RANO criteria.
Time Frame: Up to 4.1 years in Phase I and 1.4 years in Phase II
Population: as for outcome 12
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W | Phase II: BLZ945 1200 mg 4d on/10d Off QD | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 4 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 3 | 1 | 0 | 2 | 22 | 21
percentage of participants |  |  |  |  |  |  | 0 [0.0 to 95.0] |  | 0 [0.0 to 95.0] |  | 33.3 [1.7 to 86.5] |  | 50.0 [9.8 to 90.2] | 33.3 [1.7 to 86.5] |  |  |  |  | 0 [0.0 to 95.0] | 100 [5.0 to 100] | 40.0 [7.6 to 81.1] | 0 [0.0 to 63.2] | 0 [0.0 to 95.0] |  | 0 [0.0 to 77.6] | 27.3 [12.6 to 46.9] | 23.8 [9.9 to 43.7]

25. Secondary Outcome: Phase I and II: Disease Control Rate (DCR) Per iRANO
Description: DCR is the percentage of patients with a best overall response of complete response (CR), partial response (PR) or stable disease (SD), based on local investigator assessment per iRANO criteria.
Time Frame: Up to 4.1 years in Phase I and 1.4 years in Phase II
Population: as for outcome 12
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W | Phase II: BLZ945 1200 mg 4d on/10d Off QD | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 4 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 3 | 1 | 0 | 2 | 22 | 21
percentage of participants |  |  |  |  |  |  | 0 [0.0 to 95.0] |  | 0 [0.0 to 95.0] |  | 33.3 [1.7 to 86.5] |  | 50.0 [9.8 to 90.2] | 33.3 [1.7 to 86.5] |  |  |  |  | 0 [0.0 to 95.0] | 100 [5.0 to 100.0] | 40.0 [7.6 to 81.1] | 0 [0.0 to 63.2] | 0 [0.0 to 95.0] |  | 0 [0.0 to 77.6] | 27.3 [12.6 to 46.9] | 23.8 [9.9 to 43.7]

26. Secondary Outcome: Phase I: Disease Control Rate (DCR) Per Guidelines for Efficacy Evaluation in Lymphoma Studies
Description: DCR is the percentage of patients with a best overall response of complete response (CR), partial response (PR) or stable disease (SD), based on local investigator assessment per guidelines for efficacy evaluation in lymphoma studies.
Time Frame: Up to 3.1 years for BLZ945 single agent and 4.1 years for BLZ945 in combination with PDR001
Population: as for outcome 13
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
percentage of participants |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0 [0.0 to 77.6] |  |  |  |  | 50.0 [2.5 to 97.5] |  |  |

27. Secondary Outcome: Phase II: Duration of Response (DOR) Per RANO
Description: DOR only applies to patients for whom best overall response is complete response (CR) or partial response (PR) based on local investigator assessment per RANO. DOR is defined as the time from the date of first documented response to the date of first documented progression or death due to underlying cancer. If a patient did not have an event, DOR was censored at the date of last adequate tumor assessment.
Time Frame: Up to 1.4 years for BLZ945 single agent and 0.6 years for BLZ945 in combination with PDR001
Population: All patients from Phase II for whom best overall response is complete response (CR) or partial response (PR) per RANO
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: BLZ945 1200 mg 4d on/10d Off QD | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W
Number analyzed (Participants) | 3 | 0
months | 7.3 [6.7 to NA] — Not estimable due to insufficient number of participants with events. |

28. Secondary Outcome: Phase II: Duration of Response (DOR) Per iRANO
Description: DOR only applies to patients for whom best overall response is complete response (CR) or partial response (PR) based on local investigator assessment per iRANO. DOR is defined as the time from the date of first documented response to the date of first documented progression or death due to underlying cancer. If a patient did not have an event, DOR was censored at the date of last adequate tumor assessment.
Time Frame: Up to 1.4 years for BLZ945 single agent and 0.6 years for BLZ945 in combination with PDR001
Population: All patients from Phase II for whom best overall response is complete response (CR) or partial response (PR) per iRANO
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: BLZ945 1200 mg 4d on/10d Off QD | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W
Number analyzed (Participants) | 3 | 0
months | 16.2 [6.7 to NA] — Not estimable due to insufficient number of participants with events. |

29. Secondary Outcome: Phase II: Overall Survival (OS)
Description: OS is defined as the time from date of start of treatment to date of death due to any cause. If a patient was not known to have died, OS time was censored at the date of last contact.
  OS was estimated using Kaplan-Meier estimates.
Time Frame: From start of treatment until death due to any cause, assessed up to 1.9 years for BLZ945 single agent and 1.3 years for BLZ945 in combination with PDR001
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: BLZ945 1200 mg 4d on/10d Off QD | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W
Number analyzed (Participants) | 22 | 21
months | 8.4 [6.4 to 13.7] | 7.0 [2.3 to 10.9]

30. Secondary Outcome: Phase II: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) During the On-treatment Period
Description: as for outcome 1
Time Frame: From first dose of study medication up to 30 days after last dose, with a maximum duration of 1.4 years for BLZ945 single agent and 0.6 years for BLZ945 in combination with PDR001
Population: All patients from Phase II who received at least one dose of BLZ945 or PDR001. Patients were analyzed according to the study treatment (regimen) they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: BLZ945 1200 mg 4d on/10d Off QD | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W
Number analyzed (Participants) | 22 | 21
Participants
  AEs | 22 | 20
  Treatment-related AEs | 14 | 14
  SAEs | 10 | 10
  Treatment-related SAEs | 2 | 4
  Fatal SAEs | 0 | 1

31. Secondary Outcome: Phase II: Number of Participants With Dose Reductions and Dose Interruptions of BLZ945
Description: as for outcome 2
Time Frame: From first dose of study medication up to last dose, with a maximum duration of 1.3 years for BLZ945 single agent and 0.5 years for BLZ945 in combination with PDR001
Population: All patients from Phase II who received at least one dose of BLZ945. Patients were analyzed according to the study treatment (regimen) they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: BLZ945 1200 mg 4d on/10d Off QD | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W
Number analyzed (Participants) | 22 | 21
Participants
  At least one dose reduction | 1 | 1
  At least one dose interruption | 7 | 5

32. Secondary Outcome: Phase II: Number of Participants With Dose Reductions and Dose Interruptions of PDR001
Description: as for outcome 3
Time Frame: From first dose of study medication up to last dose, with a maximum duration of 0.5 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: BLZ945 1200 mg 4d on/10d Off QD | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W
Number analyzed (Participants) | 0 | 21
Participants
  At least one dose reduction |  | 0
  At least one dose interruption |  | 1

33. Secondary Outcome: Phase II: Dose Intensity of BLZ945
Description: Dose intensity of BLZ945 was calculated as cumulative actual dose in milligrams divided by the number of dose days scheduled per protocol during the treatment period. The denominator was calculated considering that patients received doses 4 days out of every 14 in the 4 days on/10 days off regimen.
Time Frame: as for outcome 31
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Phase II: BLZ945 1200 mg 4d on/10d Off QD | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W
Number analyzed (Participants) | 22 | 21
mg/day | 1104.7 (119.63) | 610.4 (83.00)

34. Secondary Outcome: Phase II: Dose Intensity of PDR001
Description: as for outcome 5
Time Frame: From first dose of study medication up to last dose, with a maximum duration of 0.5 years
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Phase II: BLZ945 1200 mg 4d on/10d Off QD | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W
Number analyzed (Participants) | 0 | 21
mg/day |  | 395.2 (21.82)

35. Secondary Outcome: Phase I and II: Maximum Observed Serum Concentration (Cmax) of BLZ945 (7d on/7d Off Regimen)
Description: Pharmacokinetic (PK) parameters were calculated based on BLZ945 serum concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed serum concentration following a dose.
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 7 (1 cycle=28 days): pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post dose
Population: Patients in the pharmacokinetic analysis set (PAS) who received BLZ945 (7d on/7d off regimen) and had an available value for the outcome measure at each timepoint. PAS consists of all patients who received one of the planned treatments, provided at least one primary PK parameter and did not vomit within 4 hours after dosing with BLZ495.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD
Number analyzed (Participants) | 5 | 7
µg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 7
  Cycle 1 Day 1 | 4.48 (1.42) | 9.33 (2.8)
  Cycle 1 Day 7: number analyzed (Participants) | 5 | 5
  Cycle 1 Day 7 | 6.58 (2.07) | 13.9 (4.51)

36. Secondary Outcome: Phase I and II: Maximum Observed Serum Concentration (Cmax) of BLZ945 (Q1W Regimen)
Description: as for outcome 35
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 8 (1 cycle=28 days): pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post dose (QD dosing); pre-dose, 0.5, 1, 2, 4, 6, 8 and 12 hours post morning dose (and pre evening dose) and 12 hours post evening dose (BID dosing)
Population: Patients in the pharmacokinetic analysis set (PAS) who received BLZ945 (Q1W regimen) and had an available value for the outcome measure at each timepoint. PAS consists of all patients who received one of the planned treatments, provided at least one primary PK parameter and did not vomit within 4 hours after dosing with BLZ495.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 5 | 6 | 3 | 5 | 6 | 0 | 3 | 4 | 5 | 8 | 5 | 6 | 5 | 3
µg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 5 | 3 | 3 | 5 | 0 | 3 | 4 | 5 | 8 | 5 | 6 | 5 | 3
  Cycle 1 Day 1 | 8.39 (1.39) | 15.4 (3.04) | 13 (3.42) | 20.1 (3.07) | 26.4 (6.42) |  | 15 (3.04) | 3.94 (0.847) | 9.02 (2.14) | 16.5 (2.97) | 18.9 (2.09) | 25.3 (4.84) | 15.5 (3.13) | 17.6 (3.12)
  Cycle 1 Day 8: number analyzed (Participants) | 4 | 6 | 3 | 5 | 6 | 0 | 3 | 3 | 5 | 8 | 5 | 5 | 5 | 3
  Cycle 1 Day 8 | 8.74 (1.84) | 13.2 (4.81) | 15.8 (3.18) | 27.1 (3.3) | 29.6 (7.22) |  | 13.6 (3.64) | 4.68 (0.731) | 9.05 (2.94) | 17.3 (2.44) | 20.6 (4.89) | 33.9 (6.92) | 16.4 (3.83) | 16.4 (3.66)

37. Secondary Outcome: Phase I and II: Maximum Observed Serum Concentration (Cmax) of BLZ945 (4d on/10d Off Regimen)
Description: as for outcome 35
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 4 (1 cycle=28 days): pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post dose (QD dosing); pre-dose, 0.5, 1, 2, 4, 6, 8 and 12 hours post morning dose (and pre evening dose) and 12 hours post evening dose (BID dosing)
Population: Patients in the pharmacokinetic analysis set (PAS) who received BLZ945 (4d on/10d off regimen) and had an available value for the outcome measure at each timepoint. PAS consists of all patients who received one of the planned treatments, provided at least one primary PK parameter and did not vomit within 4 hours after dosing with BLZ495. Patients treated at the same dose level and regimen are pooled together.
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Phase I and II: BLZ945 1200 mg 4d on/10d Off QD: BLZ945 1200 mg once per day administered for 4 days and suspended for 10 days. Patients from phase I and II treated at the same dose level and regimen pooled.
- Phase I and II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W: BLZ945 700 mg once per day administered for 4 days and suspended for 10 days in combination with PDR001 400 mg every 4 weeks. Patients from phase I and II treated at the same dose level and regimen pooled.
Arm/Group | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I and II: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I and II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W
Number analyzed (Participants) | 8 | 8 | 5 | 30 | 6 | 5 | 11 | 27 | 4
µg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 8 | 8 | 4 | 30 | 6 | 5 | 11 | 27 | 4
  Cycle 1 Day 1 | 9.59 (2.86) | 18.2 (3.44) | 16.2 (5.15) | 24.5 (5.79) | 16.5 (3.06) | 9.31 (3.47) | 11.8 (3.35) | 16.7 (4.45) | 25 (5.4)
  Cycle 1 Day 4: number analyzed (Participants) | 8 | 8 | 5 | 26 | 6 | 5 | 11 | 26 | 3
  Cycle 1 Day 4 | 14.4 (4.4) | 28.1 (4.26) | 23.6 (6.78) | 38.2 (10.1) | 30.5 (5.65) | 14.1 (3.29) | 19.3 (7.53) | 26 (8.54) | 40.3 (11.9)

38. Secondary Outcome: Phase I and II: Time to Reach Maximum Serum Concentration (Tmax) of BLZ945 (7d on/7d Off Regimen)
Description: Pharmacokinetic (PK) parameters were calculated based on BLZ945 serum concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) serum concentration following a dose. Actual recorded sampling times were considered for the calculations.
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 7 (1 cycle=28 days): pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post dose
Population: as for outcome 35
Measure: Median (Full Range); unit: hours
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD
Number analyzed (Participants) | 5 | 7
hours
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 7
  Cycle 1 Day 1 | 1.29 [0.5 to 2] | 1.88 [0.5 to 6]
  Cycle 1 Day 7: number analyzed (Participants) | 5 | 5
  Cycle 1 Day 7 | 1 [0.5 to 2] | 2.03 [1.1 to 4]

39. Secondary Outcome: Phase I and II: Time to Reach Maximum Serum Concentration (Tmax) of BLZ945 (Q1W Regimen)
Description: as for outcome 38
Time Frame: as for outcome 36
Population: as for outcome 36
Measure: Median (Full Range); unit: hours
Arm/Group | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 5 | 6 | 3 | 5 | 6 | 0 | 3 | 4 | 5 | 8 | 5 | 6 | 5 | 3
hours
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 5 | 3 | 3 | 5 | 0 | 3 | 4 | 5 | 8 | 5 | 6 | 5 | 3
  Cycle 1 Day 1 | 2.03 [1.02 to 3.92] | 1.9 [1 to 2.05] | 3.83 [2 to 4] | 2.07 [2.07 to 3.92] | 3.82 [2 to 6.13] |  | 2.17 [1.02 to 4.13] | 1.43 [0.533 to 1.95] | 1.17 [1 to 3.88] | 1.78 [0.5 to 4.37] | 2.1 [1.57 to 8] | 2.43 [1.48 to 4] | 1.88 [1.55 to 11] | 1.8 [1.6 to 4.15]
  Cycle 1 Day 8: number analyzed (Participants) | 4 | 6 | 3 | 5 | 6 | 0 | 3 | 3 | 5 | 8 | 5 | 5 | 5 | 3
  Cycle 1 Day 8 | 1.88 [0.867 to 3.92] | 1.53 [0.883 to 4.23] | 2 [1.92 to 2] | 4.07 [1.95 to 7.35] | 3 [2 to 7.05] |  | 2.12 [1.85 to 3.95] | 1.9 [1.08 to 2.13] | 1.03 [0.5 to 1.95] | 1.98 [0.5 to 4] | 1.02 [0.5 to 2.12] | 2.07 [1 to 6] | 2.05 [0.883 to 4] | 7.1 [2 to 10]

40. Secondary Outcome: Phase I and II: Time to Reach Maximum Serum Concentration (Tmax) of BLZ945 (4d on/10d Off Regimen)
Description: as for outcome 38
Time Frame: as for outcome 37
Population: as for outcome 37
Measure: Median (Full Range); unit: hours
Arm/Group | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I and II: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I and II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W
Number analyzed (Participants) | 8 | 8 | 5 | 30 | 6 | 5 | 11 | 27 | 4
hours
  Cycle 1 Day 1: number analyzed (Participants) | 8 | 8 | 4 | 30 | 6 | 5 | 11 | 27 | 4
  Cycle 1 Day 1 | 1.54 [1.03 to 2.05] | 2 [0.6 to 25.4] | 2.07 [1.22 to 6] | 2.06 [0.483 to 6.2] | 0.933 [0.567 to 3.97] | 1.95 [1 to 25.6] | 2 [0.5 to 5.83] | 2 [0.5 to 24.4] | 3 [1.23 to 5.12]
  Cycle 1 Day 4: number analyzed (Participants) | 8 | 8 | 5 | 26 | 6 | 5 | 11 | 26 | 3
  Cycle 1 Day 4 | 1.05 [0.983 to 2.02] | 2.03 [0.883 to 4.05] | 4 [2.08 to 7] | 2.04 [0.5 to 23.9] | 1.93 [1.18 to 5.85] | 2.02 [1.08 to 3.95] | 1.95 [1 to 27.9] | 1.92 [0.5 to 7] | 4 [3.88 to 6.13]

41. Secondary Outcome: Phase I and II: Area Under the Serum Concentration-time Curve From Time Zero to 24 Hours Post Dose (AUC0-24hr) of BLZ945 (7d on/7d Off Regimen)
Description: PK parameters were calculated based on BLZ945 serum concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUC0-24hr calculation.
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 7 (1 cycle=28 days): pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post dose
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: hr*µg/mL
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD
Number analyzed (Participants) | 5 | 6
hr*µg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 6
  Cycle 1 Day 1 | 56.2 (9.43) | 125 (30.8)
  Cycle 1 Day 7: number analyzed (Participants) | 5 | 4
  Cycle 1 Day 7 | 89.8 (35.9) | 226 (72.1)

42. Secondary Outcome: Phase I and II: Area Under the Serum Concentration-time Curve From Time Zero to 24 Hours Post Dose (AUC0-24hr) of BLZ945 (Q1W Regimen, QD Dosing)
Description: as for outcome 41
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 8 (1 cycle=28 days): pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post dose
Population: Patients in the pharmacokinetic analysis set (PAS) who received BLZ945 (Q1W regimen, QD dosing) and had an available value for the outcome measure at each timepoint. PAS consists of all patients who received one of the planned treatments, provided at least one primary PK parameter and did not vomit within 4 hours after dosing with BLZ495.
Measure: Mean (Standard Deviation); unit: hr*µg/mL
Arm/Group | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 5 | 6 | 3 | 3 | 6 | 0 | 0 | 4 | 5 | 8 | 5 | 6 | 0 | 0
hr*µg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 5 | 3 | 3 | 4 | 0 | 0 | 4 | 5 | 7 | 4 | 6 | 0 | 0
  Cycle 1 Day 1 | 118 (17.3) | 187 (43.3) | 211 (44.1) | 326 (39.9) | 399 (48.1) |  |  | 51.6 (20.8) | 118 (27) | 218 (19.5) | 290 (20.5) | 410 (76) |  |
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 6 | 3 | 3 | 6 | 0 | 0 | 3 | 5 | 8 | 5 | 5 | 0 | 0
  Cycle 1 Day 8 | 136 (31.9) | 182 (71.9) | 226 (48.5) | 422 (95) | 481 (126) |  |  | 69.4 (8.67) | 120 (27.7) | 233 (37.3) | 323 (105) | 486 (118) |  |

43. Secondary Outcome: Phase I and II: Area Under the Serum Concentration-time Curve From Time Zero to 12 Hours Post Dose (AUC0-12hr) of BLZ945 (Q1W Regimen, BID Dosing)
Description: PK parameters were calculated based on BLZ945 serum concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUC0-12hr calculation.
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 8 (1 cycle=28 days): pre-dose, 0.5, 1, 2, 4, 6, 8 and 12 hours post morning dose (and pre evening dose) and 12 hours post evening dose
Population: Patients in the pharmacokinetic analysis set (PAS) who received BLZ945 (Q1W regimen, BID dosing) and had an available value for the outcome measure at each timepoint. PAS consists of all patients who received one of the planned treatments, provided at least one primary PK parameter and did not vomit within 4 hours after dosing with BLZ495.
Measure: Mean (Standard Deviation); unit: hr*µg/mL
Arm/Group | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 5 | 2
hr*µg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Cycle 1 Day 1 |  |  |  |  |  |  | 127 (38.8) |  |  |  |  |  | 119 (1.69) | 159 (27.2)
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1
  Cycle 1 Day 8 |  |  |  |  |  |  |  |  |  |  |  |  | 142 (30.4) | 165

44. Secondary Outcome: Phase I and II: Area Under the Serum Concentration-time Curve From Time Zero to 24 Hours Post Dose (AUC0-24hr) of BLZ945 (4d on/10d Off Regimen, QD Dosing)
Description: as for outcome 41
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 4 (1 cycle=28 days): pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post dose
Population: Patients in the pharmacokinetic analysis set (PAS) who received BLZ945 (4d on/10d off regimen, QD dosing) and had an available value for the outcome measure at each timepoint. PAS consists of all patients who received one of the planned treatments, provided at least one primary PK parameter and did not vomit within 4 hours after dosing with BLZ495. Patients treated at the same dose level and regimen are pooled together.
Measure: Mean (Standard Deviation); unit: hr*µg/mL
Arm/Group | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I and II: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I and II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W
Number analyzed (Participants) | 8 | 8 | 4 | 26 | 0 | 5 | 11 | 27 | 3
hr*µg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 8 | 8 | 4 | 26 | 0 | 5 | 10 | 27 | 3
  Cycle 1 Day 1 | 117 (26.7) | 268 (32.2) | 241 (74.2) | 371 (88.6) |  | 138 (39.2) | 165 (54.1) | 231 (62.2) | 424 (87.9)
  Cycle 1 Day 4: number analyzed (Participants) | 8 | 7 | 4 | 20 | 0 | 4 | 11 | 21 | 2
  Cycle 1 Day 4 | 212 (71.7) | 444 (88.6) | 418 (73.1) | 653 (189) |  | 197 (95.6) | 301 (124) | 431 (156) | 656 (224)

45. Secondary Outcome: Phase I and II: Area Under the Serum Concentration-time Curve From Time Zero to 12 Hours Post Dose (AUC0-12hr) of BLZ945 (4d on/10d Off Regimen, BID Dosing)
Description: as for outcome 43
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 4 (1 cycle=28 days): pre-dose, 0.5, 1, 2, 4, 6, 8 and 12 hours post morning dose (and pre evening dose) and 12 hours post evening dose
Population: Patients in the pharmacokinetic analysis set (PAS) who received BLZ945 (4d on/10d off regimen, BID dosing) and had an available value for the outcome measure at each timepoint. PAS consists of all patients who received one of the planned treatments, provided at least one primary PK parameter and did not vomit within 4 hours after dosing with BLZ495. Patients treated at the same dose level and regimen are pooled together.
Measure: Mean (Standard Deviation); unit: hr*µg/mL
Arm/Group | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I and II: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I and II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
hr*µg/mL
  Cycle 1 Day 1 |  |  |  |  | 123 (31.4) |  |  |  |
  Cycle 1 Day 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
  Cycle 1 Day 4 |  |  |  |  | 235 (51.9) |  |  |  |

46. Secondary Outcome: Phase I and II: Maximum Observed Serum Concentration (Cmax) of PDR001
Description: Pharmacokinetic (PK) parameters were calculated based on PDR001 serum concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed serum concentration following a dose.
Time Frame: pre-infusion and 1, 24, 168, 336 and 672 hours after completion of the infusion on Cycle 1 Day 1 and Cycle 3 Day 1. The average duration of the infusion was 30 minutes. The duration of one cycle was 28 days
Population: Patients in the pharmacokinetic analysis set (PAS) who received PDR001 and had an available value for the outcome measure at each timepoint. PAS consists of all patients who received one of the planned treatments, provided at least one primary PK parameter and did not vomit within 4 hours after dosing with BLZ495. Patients treated at the same dose level and regimen are pooled together.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I and II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 4 | 5 | 9 | 4 | 6 | 5 | 10 | 26 | 4 | 5 | 5
µg/mL
  Cycle 1 Day 1 | 102 (13.6) | 93.8 (26.3) | 102 (20.9) | 96.3 (25.7) | 111 (25.2) | 102 (10.5) | 102 (19.4) | 99.4 (27.6) | 122 (5.35) | 111 (25.1) | 102 (28)
  Cycle 3 Day 1: number analyzed (Participants) | 2 | 3 | 3 | 2 | 2 | 2 | 5 | 4 | 0 | 2 | 0
  Cycle 3 Day 1 | 120 (42.3) | 132 (16.1) | 142 (38.1) | 114 (40.4) | 138 (54.2) | 137 (55.4) | 156 (48.5) | 126 (55.6) |  | 118 (44.3) |

47. Secondary Outcome: Phase I and II: Time to Reach Maximum Serum Concentration (Tmax) of PDR001
Description: Pharmacokinetic (PK) parameters were calculated based on PDR001 serum concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) serum concentration following a dose. Actual recorded sampling times were considered for the calculations.
Time Frame: as for outcome 46
Population: as for outcome 46
Measure: Median (Full Range); unit: hours
Arm/Group | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I and II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 4 | 5 | 9 | 4 | 6 | 5 | 10 | 26 | 4 | 5 | 5
hours
  Cycle 1 Day 1 | 1.67 [0.833 to 24.2] | 1.45 [0.833 to 1.67] | 1.5 [0.85 to 1.67] | 1.28 [0.933 to 2.1] | 1.48 [0.983 to 24.5] | 1.42 [0.3 to 23] | 1.48 [1.03 to 23.2] | 1.79 [1 to 90.6] | 1.46 [1.28 to 23.8] | 1.53 [1.28 to 24.5] | 1.55 [1.4 to 23]
  Cycle 3 Day 1: number analyzed (Participants) | 2 | 3 | 3 | 2 | 2 | 2 | 5 | 4 | 0 | 2 | 0
  Cycle 3 Day 1 | 1.48 [1.42 to 1.55] | 1.45 [0 to 1.55] | 1.58 [1.53 to 1.65] | 1.81 [1.5 to 2.12] | 13 [2.05 to 24] | 1.53 [1.52 to 1.53] | 1.53 [1.42 to 24] | 12.7 [1.5 to 336] |  | 94.4 [1.6 to 187] |

48. Secondary Outcome: Phase I and II: Area Under the Serum Concentration-time Curve From Time Zero to 28 Days Post Dose (AUC0-28day) of PDR001
Description: PK parameters were calculated based on PDR001 serum concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUC0-28day calculation.
Time Frame: as for outcome 46
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: day*µg/mL
Arm/Group | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I and II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W
Number analyzed (Participants) | 4 | 4 | 8 | 3 | 5 | 5 | 8 | 19 | 3 | 0 | 0
day*µg/mL
  Cycle 1 Day 1 | 1390 (250) | 1120 (203) | 1160 (228) | 1130 (274) | 1310 (301) | 1350 (468) | 1270 (204) | 1230 (308) | 1330 (183) |  |
  Cycle 3 Day 1: number analyzed (Participants) | 2 | 1 | 3 | 1 | 1 | 2 | 5 | 2 | 0 | 0 | 0
  Cycle 3 Day 1 | 1960 (297) | 1780 | 1930 (630) | 1480 | 1240 | 1750 (838) | 2350 (439) | 1950 (1220) |  |  |

49. Secondary Outcome: Phase I and II: Number of Participants With Anti-PDR001 Antibodies
Description: Immunogenicity was evaluated in serum in a validated three-tiered assay approach. Samples were screened for potential anti-PDR001 antibodies and positive screen results were confirmed using a confirmatory assay. For confirmed anti-drug antibodies (ADA) positive samples, titers were determined. Patient ADA status was defined as follows:
  * ADA-negative at baseline: ADA-negative sample at baseline
  * ADA-positive at baseline: ADA-positive sample at baseline
  * ADA-negative post-baseline: patient with ADA-negative sample at baseline and at least 1 post baseline determinant sample, all of which are ADA-negative samples
  * Treatment-induced ADA-positive = ADA-negative sample at baseline and at least 1 treatment-induced ADA-positive sample
  * Treatment-boosted ADA-positive = ADA-positive sample at baseline and at least 1 treatment-boosted ADA-positive sample
Time Frame: Baseline (before first dose) and post-baseline (assessed throughout the treatment and safety follow-up, up to 4.4 years in phase I and 0.9 years in phase II).
Population: All patients who received at least one full or partial dose of the combination BLZ945+PDR001 and had a determinant baseline immunogenicity (IG) sample and at least one determinant post-baseline IG sample for assessing anti-PDR001 antibodies. Determinant samples are defined as samples which are not unevaluable (where unevaluable = sample where assay is not available).
Measure: Number; unit: participants
Arm/Group | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W
Number analyzed (Participants) | 3 | 5 | 6 | 5 | 6 | 5 | 10 | 7 | 4 | 5 | 4 | 17
participants
  ADA-negative at baseline | 3 | 5 | 5 | 4 | 6 | 4 | 10 | 7 | 4 | 5 | 4 | 17
  ADA-positive at baseline | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  ADA-negative post-baseline: number analyzed (Participants) | 3 | 5 | 5 | 4 | 6 | 4 | 10 | 7 | 4 | 5 | 4 | 17
  ADA-negative post-baseline | 3 | 5 | 4 | 4 | 6 | 4 | 8 | 7 | 4 | 5 | 4 | 17
  Treatment-induced ADA-positive: number analyzed (Participants) | 3 | 5 | 5 | 4 | 6 | 4 | 10 | 7 | 4 | 5 | 4 | 17
  Treatment-induced ADA-positive | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Treatment-boosted ADA-positive: number analyzed (Participants) | 3 | 5 | 5 | 4 | 6 | 4 | 10 | 7 | 4 | 5 | 4 | 17
  Treatment-boosted ADA-positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

50. Post Hoc Outcome: All-Collected Deaths
Description: On-treatment and post-treatment safety follow-up deaths were collected from first dose of study medication to 30 days after last dose (BLZ945 single agent; SA) and to 150 days after last dose (BLZ945+PDR001; combo). Survival follow-up deaths were collected from 31 days (SA) and 151 days (combo) after last dose until end of study. All deaths refer to the sum of on-treatment and post-treatment safety follow-up deaths plus survival follow-up deaths.
Time Frame: On&post-treatment safety: up to 3.1 years (phase I)/1.4 years (phase II) for SA and 4.4 years (phase I)/0.9 years (phase II) for combo. Survival: up to 3.1 years (phase I)/1.9 years (phase II) for SA and 4.4 years (phase I)/1.3 years (phase II) for combo
Population: All patients who received at least one dose of assigned single agent BLZ945, or at least one full or partial dose of assigned combination BLZ945+PDR001. Patients were analyzed according to the study treatment (regimen) they actually received.
Measure: Number; unit: participants
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W | Phase II: BLZ945 1200 mg 4d on/10d Off QD | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W
Number analyzed (Participants) | 5 | 7 | 5 | 6 | 3 | 5 | 6 | 8 | 9 | 5 | 10 | 1 | 4 | 6 | 4 | 5 | 9 | 5 | 6 | 5 | 11 | 9 | 4 | 6 | 5 | 22 | 21
participants
  On-treatment and post-treatment safety follow-up deaths | 1 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 4 | 3 | 3 | 3 | 2 | 6 | 4 | 3 | 4 | 2 | 2 | 8
  Survival follow-up deaths: number analyzed (Participants) | 4 | 7 | 4 | 4 | 3 | 5 | 4 | 8 | 8 | 5 | 9 | 1 | 2 | 5 | 4 | 1 | 6 | 2 | 3 | 3 | 5 | 5 | 1 | 2 | 3 | 20 | 13
  Survival follow-up deaths | 4 | 4 | 3 | 3 | 3 | 5 | 3 | 7 | 7 | 4 | 6 | 1 | 2 | 5 | 2 | 1 | 3 | 2 | 1 | 0 | 2 | 2 | 0 | 1 | 3 | 14 | 9
  All deaths | 5 | 4 | 4 | 5 | 3 | 5 | 5 | 7 | 8 | 4 | 7 | 1 | 4 | 6 | 2 | 5 | 6 | 5 | 4 | 2 | 8 | 6 | 3 | 5 | 5 | 16 | 17

ADVERSE EVENTS:
Time Frame: On-treatment and post-treatment safety follow-up: from first dose of study treatment to 30 days after last dose (single agent; SA) and to 150 days after last dose (combo), up to 3.1 years (phase I)/1.4 years (phase II) for SA and 4.4 years (phase I)/0.9 years (phase II) for combo. Deaths in survival period: from 31 days (SA) and 151 days (combo) after last dose until end of study, up to 3.1 years (phase I)/1.9 years (phase II) for SA and 4.4 years (phase I)/1.3 years (phase II) for combo.
Description: Deaths in the survival period are not considered Adverse Events (AEs). No AEs were collected in the survival period.
Groups:
- Phase I: BLZ945 150 mg 7d on/7d Off QD; Phase I: BLZ945 300 mg 7d on/7d Off QD; Phase I: BLZ945 300 mg Q1W QD; Phase I: BLZ945 450 mg Q1W QD; Phase I: BLZ945 600 mg Q1W QD; Phase I: BLZ945 1000 mg Q1W QD; Phase I: BLZ945 1600 mg Q1W QD; Phase I: BLZ945 300 mg 4d on/10d Off QD; Phase I: BLZ945 600 mg 4d on/10d Off QD; Phase I: BLZ945 800 mg 4d on/10d Off QD; Phase I: BLZ945 1200 mg 4d on/10d Off QD; Phase I: BLZ945 300 mg Q1W BID; Phase I: BLZ945 600 mg Q1W BID; Phase I: BLZ945 600 mg 4d on/10d Off BID; Phase II: BLZ945 1200 mg 4d on/10d Off QD: Safety data up to 30 days after last dose
- Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W; Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W; Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W; Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W; Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W; Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W; Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W; Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W; Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W; Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W; Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W; Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W: Safety data up to 150 days after last dose
- Phase I: BLZ945 150 mg 7d on/7d Off QD - Survival Period; Phase I: BLZ945 300 mg 7d on/7d Off QD - Survival Period; Phase I: BLZ945 300 mg Q1W QD - Survival Period; Phase I: BLZ945 450 mg Q1W QD - Survival Period; Phase I: BLZ945 600 mg Q1W QD - Survival Period; Phase I: BLZ945 1000 mg Q1W QD - Survival Period; Phase I: BLZ945 1600 mg Q1W QD - Survival Period; Phase I: BLZ945 300 mg 4d on/10d Off QD - Survival Period; Phase I: BLZ945 600 mg 4d on/10d Off QD - Survival Period; Phase I: BLZ945 800 mg 4d on/10d Off QD - Survival Period; Phase I: BLZ945 1200 mg 4d on/10d Off QD - Survival Period; Phase I: BLZ945 300 mg Q1W BID - Survival Period; Phase I: BLZ945 600 mg Q1W BID - Survival Period; Phase I: BLZ945 600 mg 4d on/10d Off BID - Survival Period; Phase II: BLZ945 1200 mg 4d on/10d Off QD - Survival Period: Deaths collected in the survival follow-up period (starting from Day 31 post-treatment for BLZ945 single agent). No AEs were collected during this period.
- Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W - Survival Period; Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W - Survival Period; Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W - Survival Period; Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W - Survival Period; Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W - Survival Period; Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W - Survival Period; Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W - Survival Period; Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W - Survival Period; Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W - Survival Period; Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W - Survival Period; Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W - Survival Period; Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W - Survival Period: Deaths collected in the survival follow-up period (starting from Day 151 post-treatment for BLZ945+PDR001). No AEs were collected during this period.
Arm/Group | Phase I: BLZ945 150 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg 7d on/7d Off QD | Phase I: BLZ945 300 mg Q1W QD | Phase I: BLZ945 450 mg Q1W QD | Phase I: BLZ945 600 mg Q1W QD | Phase I: BLZ945 1000 mg Q1W QD | Phase I: BLZ945 1600 mg Q1W QD | Phase I: BLZ945 300 mg 4d on/10d Off QD | Phase I: BLZ945 600 mg 4d on/10d Off QD | Phase I: BLZ945 800 mg 4d on/10d Off QD | Phase I: BLZ945 1200 mg 4d on/10d Off QD | Phase I: BLZ945 300 mg Q1W BID | Phase I: BLZ945 600 mg Q1W BID | Phase I: BLZ945 600 mg 4d on/10d Off BID | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W | Phase II: BLZ945 1200 mg 4d on/10d Off QD | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W | Phase I: BLZ945 150 mg 7d on/7d Off QD - Survival Period | Phase I: BLZ945 300 mg 7d on/7d Off QD - Survival Period | Phase I: BLZ945 300 mg Q1W QD - Survival Period | Phase I: BLZ945 450 mg Q1W QD - Survival Period | Phase I: BLZ945 600 mg Q1W QD - Survival Period | Phase I: BLZ945 1000 mg Q1W QD - Survival Period | Phase I: BLZ945 1600 mg Q1W QD - Survival Period | Phase I: BLZ945 300 mg 4d on/10d Off QD - Survival Period | Phase I: BLZ945 600 mg 4d on/10d Off QD - Survival Period | Phase I: BLZ945 800 mg 4d on/10d Off QD - Survival Period | Phase I: BLZ945 1200 mg 4d on/10d Off QD - Survival Period | Phase I: BLZ945 300 mg Q1W BID - Survival Period | Phase I: BLZ945 600 mg Q1W BID - Survival Period | Phase I: BLZ945 600 mg 4d on/10d Off BID - Survival Period | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W - Survival Period | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W - Survival Period | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W - Survival Period | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W - Survival Period | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W - Survival Period | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W - Survival Period | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W - Survival Period | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W - Survival Period | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W - Survival Period | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W - Survival Period | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W - Survival Period | Phase II: BLZ945 1200 mg 4d on/10d Off QD - Survival Period | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W - Survival Period
All-Cause Mortality (participants affected / at risk) | 1/5 | 0/7 | 1/5 | 2/6 | 0/3 | 0/5 | 2/6 | 0/8 | 1/9 | 0/5 | 1/10 | 0/1 | 2/4 | 1/6 | 0/4 | 4/5 | 3/9 | 3/5 | 3/6 | 2/5 | 6/11 | 4/9 | 3/4 | 4/6 | 2/5 | 2/22 | 8/21 | 4/4 | 4/7 | 3/4 | 3/4 | 3/3 | 5/5 | 3/4 | 7/8 | 7/8 | 4/5 | 6/9 | 1/1 | 2/2 | 5/5 | 2/4 | 1/1 | 3/6 | 2/2 | 1/3 | 0/3 | 2/5 | 2/5 | 0/1 | 1/2 | 3/3 | 14/20 | 9/13
Serious Adverse Events (participants affected / at risk) | 3/5 | 1/7 | 3/5 | 2/6 | 0/3 | 3/5 | 3/6 | 4/8 | 3/9 | 3/5 | 5/10 | 0/1 | 3/4 | 5/6 | 1/4 | 2/5 | 6/9 | 4/5 | 3/6 | 1/5 | 6/11 | 7/9 | 4/4 | 2/6 | 1/5 | 10/22 | 11/21 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 5/5 | 7/7 | 5/5 | 6/6 | 3/3 | 5/5 | 6/6 | 8/8 | 9/9 | 5/5 | 10/10 | 1/1 | 4/4 | 6/6 | 4/4 | 5/5 | 9/9 | 5/5 | 6/6 | 5/5 | 11/11 | 9/9 | 4/4 | 6/6 | 5/5 | 20/22 | 19/21 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: BLZ945 150 mg 7d on/7d Off QD (N=5) | Phase I: BLZ945 300 mg 7d on/7d Off QD (N=7) | Phase I: BLZ945 300 mg Q1W QD (N=5) | Phase I: BLZ945 450 mg Q1W QD (N=6) | Phase I: BLZ945 600 mg Q1W QD (N=3) | Phase I: BLZ945 1000 mg Q1W QD (N=5) | Phase I: BLZ945 1600 mg Q1W QD (N=6) | Phase I: BLZ945 300 mg 4d on/10d Off QD (N=8) | Phase I: BLZ945 600 mg 4d on/10d Off QD (N=9) | Phase I: BLZ945 800 mg 4d on/10d Off QD (N=5) | Phase I: BLZ945 1200 mg 4d on/10d Off QD (N=10) | Phase I: BLZ945 300 mg Q1W BID (N=1) | Phase I: BLZ945 600 mg Q1W BID (N=4) | Phase I: BLZ945 600 mg 4d on/10d Off BID (N=6) | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W (N=4) | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W (N=5) | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W (N=9) | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W (N=5) | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W (N=6) | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W (N=5) | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W (N=11) | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W (N=9) | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W (N=4) | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W (N=6) | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W (N=5) | Phase II: BLZ945 1200 mg 4d on/10d Off QD (N=22) | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W (N=21) | Phase I: BLZ945 150 mg 7d on/7d Off QD - Survival Period (N=0) | Phase I: BLZ945 300 mg 7d on/7d Off QD - Survival Period (N=0) | Phase I: BLZ945 300 mg Q1W QD - Survival Period (N=0) | Phase I: BLZ945 450 mg Q1W QD - Survival Period (N=0) | Phase I: BLZ945 600 mg Q1W QD - Survival Period (N=0) | Phase I: BLZ945 1000 mg Q1W QD - Survival Period (N=0) | Phase I: BLZ945 1600 mg Q1W QD - Survival Period (N=0) | Phase I: BLZ945 300 mg 4d on/10d Off QD - Survival Period (N=0) | Phase I: BLZ945 600 mg 4d on/10d Off QD - Survival Period (N=0) | Phase I: BLZ945 800 mg 4d on/10d Off QD - Survival Period (N=0) | Phase I: BLZ945 1200 mg 4d on/10d Off QD - Survival Period (N=0) | Phase I: BLZ945 300 mg Q1W BID - Survival Period (N=0) | Phase I: BLZ945 600 mg Q1W BID - Survival Period (N=0) | Phase I: BLZ945 600 mg 4d on/10d Off BID - Survival Period (N=0) | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W - Survival Period (N=0) | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W - Survival Period (N=0) | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W - Survival Period (N=0) | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W - Survival Period (N=0) | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W - Survival Period (N=0) | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W - Survival Period (N=0) | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W - Survival Period (N=0) | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W - Survival Period (N=0) | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W - Survival Period (N=0) | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W - Survival Period (N=0) | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W - Survival Period (N=0) | Phase II: BLZ945 1200 mg 4d on/10d Off QD - Survival Period (N=0) | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W - Survival Period (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cerebral palsy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal wall haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haemoperitoneum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Condition aggravated (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sudden death (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Brain herniation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Autoimmune arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cutaneous T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Peritumoural oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Brain oedema (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neurological decompensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Nephrostomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypertensive urgency (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: BLZ945 150 mg 7d on/7d Off QD (N=5) | Phase I: BLZ945 300 mg 7d on/7d Off QD (N=7) | Phase I: BLZ945 300 mg Q1W QD (N=5) | Phase I: BLZ945 450 mg Q1W QD (N=6) | Phase I: BLZ945 600 mg Q1W QD (N=3) | Phase I: BLZ945 1000 mg Q1W QD (N=5) | Phase I: BLZ945 1600 mg Q1W QD (N=6) | Phase I: BLZ945 300 mg 4d on/10d Off QD (N=8) | Phase I: BLZ945 600 mg 4d on/10d Off QD (N=9) | Phase I: BLZ945 800 mg 4d on/10d Off QD (N=5) | Phase I: BLZ945 1200 mg 4d on/10d Off QD (N=10) | Phase I: BLZ945 300 mg Q1W BID (N=1) | Phase I: BLZ945 600 mg Q1W BID (N=4) | Phase I: BLZ945 600 mg 4d on/10d Off BID (N=6) | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W (N=4) | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W (N=5) | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W (N=9) | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W (N=5) | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W (N=6) | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W (N=5) | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W (N=11) | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W (N=9) | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W (N=4) | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W (N=6) | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W (N=5) | Phase II: BLZ945 1200 mg 4d on/10d Off QD (N=22) | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W (N=21) | Phase I: BLZ945 150 mg 7d on/7d Off QD - Survival Period (N=0) | Phase I: BLZ945 300 mg 7d on/7d Off QD - Survival Period (N=0) | Phase I: BLZ945 300 mg Q1W QD - Survival Period (N=0) | Phase I: BLZ945 450 mg Q1W QD - Survival Period (N=0) | Phase I: BLZ945 600 mg Q1W QD - Survival Period (N=0) | Phase I: BLZ945 1000 mg Q1W QD - Survival Period (N=0) | Phase I: BLZ945 1600 mg Q1W QD - Survival Period (N=0) | Phase I: BLZ945 300 mg 4d on/10d Off QD - Survival Period (N=0) | Phase I: BLZ945 600 mg 4d on/10d Off QD - Survival Period (N=0) | Phase I: BLZ945 800 mg 4d on/10d Off QD - Survival Period (N=0) | Phase I: BLZ945 1200 mg 4d on/10d Off QD - Survival Period (N=0) | Phase I: BLZ945 300 mg Q1W BID - Survival Period (N=0) | Phase I: BLZ945 600 mg Q1W BID - Survival Period (N=0) | Phase I: BLZ945 600 mg 4d on/10d Off BID - Survival Period (N=0) | Phase I: BLZ945 150 mg Q1W QD + PDR001 400 mg Q4W - Survival Period (N=0) | Phase I: BLZ945 300 mg Q1W QD + PDR001 400 mg Q4W - Survival Period (N=0) | Phase I: BLZ945 600 mg Q1W QD + PDR001 400 mg Q4W - Survival Period (N=0) | Phase I: BLZ945 1000 mg Q1W QD + PDR001 400 mg Q4W - Survival Period (N=0) | Phase I: BLZ945 1400 mg Q1W QD + PDR001 400 mg Q4W - Survival Period (N=0) | Phase I: BLZ945 300 mg 4d on/10d Off QD + PDR001 400 mg Q4W - Survival Period (N=0) | Phase I: BLZ945 450 mg 4d on/10d Off QD + PDR001 400 mg Q4W - Survival Period (N=0) | Phase I: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W - Survival Period (N=0) | Phase I: BLZ945 1200 mg 4d on/10d Off QD + PDR001 400 mg Q4W - Survival Period (N=0) | Phase I: BLZ945 600 mg Q1W BID + PDR001 400 mg Q4W - Survival Period (N=0) | Phase I: BLZ945 800 mg Q1W BID + PDR001 400 mg Q4W - Survival Period (N=0) | Phase II: BLZ945 1200 mg 4d on/10d Off QD - Survival Period (N=0) | Phase II: BLZ945 700 mg 4d on/10d Off QD + PDR001 400 mg Q4W - Survival Period (N=0)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 1 | 1 | 0 | 4 | 1 | 2 | 1 | 0 | 4 | 0 | 1 | 3 | 0 | 2 | 3 | 1 | 3 | 1 | 4 | 3 | 0 | 2 | 2 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypergammaglobulinaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Diplopia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Exophthalmos (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Orbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Periorbital oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Periorbital swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Swelling of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 1 | 2 | 0 | 1 | 1 | 1 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 3 | 0 | 0 | 2 | 0 | 3 | 0 | 1 | 2 | 1 | 2 | 4 | 0 | 2 | 0 | 1 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 1 | 4 | 3 | 2 | 6 | 3 | 5 | 0 | 1 | 3 | 0 | 1 | 2 | 3 | 5 | 1 | 4 | 3 | 2 | 2 | 3 | 9 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rectal tenesmus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tongue discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 0 | 4 | 4 | 4 | 2 | 3 | 2 | 0 | 1 | 4 | 1 | 1 | 1 | 1 | 4 | 2 | 4 | 3 | 2 | 3 | 3 | 6 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Administration site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Asthenia (General disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 6 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Fatigue (General disorders) | 2 | 1 | 2 | 2 | 2 | 2 | 1 | 0 | 1 | 2 | 2 | 0 | 2 | 2 | 1 | 2 | 2 | 2 | 0 | 2 | 4 | 4 | 0 | 2 | 4 | 7 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Feeling jittery (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oedema peripheral (General disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pyrexia (General disorders) | 5 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 4 | 3 | 1 | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 2 | 1 | 3 | 1 | 2 | 1 | 2 | 3 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Swelling face (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Xerosis (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Deficiency of bile secretion (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Contrast media allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pilonidal disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Postoperative abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pyuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Breast injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 0 | 3 | 4 | 0 | 0 | 1 | 1 | 3 | 3 | 0 | 1 | 0 | 1 | 3 | 1 | 1 | 3 | 2 | 1 | 2 | 7 | 1 | 3 | 2 | 3 | 3 | 11 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Amylase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Amylase increased (Investigations) | 0 | 3 | 0 | 0 | 0 | 2 | 1 | 4 | 3 | 0 | 2 | 0 | 1 | 3 | 0 | 1 | 1 | 1 | 1 | 1 | 4 | 2 | 2 | 0 | 0 | 5 | 9 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Aspartate aminotransferase (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Aspartate aminotransferase decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 1 | 5 | 4 | 1 | 2 | 3 | 3 | 4 | 5 | 2 | 5 | 0 | 2 | 3 | 1 | 0 | 5 | 4 | 3 | 3 | 7 | 2 | 2 | 3 | 4 | 4 | 12 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood chloride decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood chloride increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood creatine phosphokinase increased (Investigations) | 0 | 3 | 0 | 2 | 0 | 1 | 3 | 3 | 5 | 0 | 3 | 0 | 1 | 2 | 0 | 0 | 3 | 3 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 8 | 7 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood creatinine (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood sodium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lipase increased (Investigations) | 1 | 2 | 0 | 0 | 1 | 2 | 0 | 3 | 3 | 0 | 1 | 0 | 3 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 2 | 6 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 3 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Troponin I increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Troponin T increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Weight decreased (Investigations) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3 | 2 | 1 | 1 | 0 | 1 | 0 | 3 | 2 | 2 | 0 | 0 | 2 | 1 | 2 | 2 | 1 | 2 | 3 | 3 | 2 | 1 | 1 | 2 | 2 | 4 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Steroid diabetes (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cancer fatigue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Agnosia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 3 | 2 | 0 | 1 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gait apraxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Headache (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 6 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hemiplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neurological decompensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neurological symptom (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Slow speech (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Bradyphrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Euphoric mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 3 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Choluria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Breast inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Nipple pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rectocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 2 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 3 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 2 | 1 | 2 | 4 | 1 | 2 | 0 | 1 | 4 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Thrombophlebitis migrans (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT02829723/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/23/NCT02829723/SAP_001.pdf